CLINICAL TRIAL: NCT02974010
Title: Sequential Therapy (NRX-100 Followed by NRX-101) for the Treatment of Acute Suicidal Ideation and Behavior in Bipolar Depression: the STABIL-B Study
Brief Title: Sequential Therapy for the Treatment of Severe Bipolar Depression.
Acronym: STABIL-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroRx, Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other); Target Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRX 101-001
Record Dates: First submitted 2016-11-22; First posted 2016-11-28 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Bipolar Depression; Suicidal Ideas; Suicidal Ideation; Suicide, Attempted
Keywords: d-cycloserine; lurasidone; ketamine; randomized controlled trial
MeSH Terms: conditions — Bipolar Disorder; Suicidal Ideation; Suicide, Attempted | interventions — Cycloserine; Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NRX-101 (Experimental): NRX-101 is a fixed dose combination of d-cycloserine and lurasidone
  Interventions: Drug: NRX-101 Oral Capsule; Drug: Ketamine Intravenous Infusion; Drug: Saline Solution Intravenous Infusion
- Lurasidone (Active Comparator): Lurasidone will be administered in the same dosages as the lurasidone component of NRX-101
  Interventions: Drug: Lurasidone Oral Capsule; Drug: Ketamine Intravenous Infusion; Drug: Saline Solution Intravenous Infusion

INTERVENTIONS:
Drug: NRX-101 Oral Capsule — Prospective Randomized Factorial Design Study as per arm/group descriptions
  Other Names: D-cycloserine + Lurasidone Fixed Dose Combination
  Arms: NRX-101
Drug: Lurasidone Oral Capsule — Prospective Randomized Factorial Design Study as per arm/group descriptions
  Other Names: Lurasidone Fixed Dose Combination
  Arms: Lurasidone
Drug: Ketamine Intravenous Infusion — Randomized administration of Ketamine or Placebo in a 3 to 1 ratio
Drug: Saline Solution Intravenous Infusion — Randomized administration of Ketamine or Placebo in a 3 to 1 ratio

SUMMARY:
NeuroRx is developing NRX-101, a fixed-dose combination oral capsule composed of d-cycloserine (DCS) and lurasidone for the maintenance of remission from Severe Bipolar Depression with Acute Suicidal Ideation (C-SSRS level 4 or 5) or Behavior (ASIB) in following initial stabilization. Patients with Severe Bipolar Depression and ASIB will be recruited in both inpatient and outpatient settings and, following informed consent, will be given an intravenous infusion of ketamine 0.5mg/kg over 40 minutes. Those who exhibit a satisfactory clinical response to ketamine will be randomly allocated to NRX-101 or to lurasidone alone (the comparator group). This study is conducted as a feasibility study for a pivotal phase 2b/3 clinical trial and the primary outcomes for this phase 2 study were blood levels of NRX-101, in order to confirm pharmaco-kinetics with remission from depression, as measured by BISS-derived MADRS and relapse as secondary outcomes.

DETAILED DESCRIPTION:
NeuroRx is developing NRX-101, a fixed-dose combination oral capsule composed of D-cycloserine (DCS) and lurasidone for the maintenance of remission from Severe Bipolar Depression with Acute Suicidal Ideation or Behavior (ASIB) in adults with Bipolar Depression following initial stabilization with ketamine. In recent years, intravenous and intranasal ketamine have demonstrated rapid and potent effects in achieving remission from both depression and suicidal ideation in both bipolar depression and major depressive disorder. However ketamine is will understood to induce hallucination and other dissociative side effects, to be addictive and have high abuse potential, and to have potential neurotoxic effects. Moreover, ketamine can only be administered in a monitored hospital or clinic setting. NRX-101 was developed with the objective of seeking a safe, non-hallucinogenic, non-addictive, oral medication that might maintain the effects of ketamine in patients with severe depression and acute suicidal ideation and which might be considered as initial therapy for patients with depression and non-acute suicidal ideation. The D-cycloserine component of NRX-101 is believed to act by inhibiting the brain's NMDA receptor and raising levels of glutamate/glutamine (Glx) in the anterior cingulate cortex. Increased Glx, as measured by magnetic resonance spectroscopy, has been associated with clinical improvement following electroconvulsive therapy (ECT) and following administration of IV ketamine.

The proposed oral combination product is intended to be administered as part of a sequential therapy consisting of the following 2 components:

1. an initial, one-time intravenous (iv) infusion of ketamine (0.5 mg/kg administered over 40 min), followed one day later by
2. twice daily oral capsules of NRX 101 (DCS + lurasidone), dosing of which is initiated 1 day after ketamine administration, titrated over 5 days to a maintenance dose and continued for up to 6 weeks. Each NRX-101 oral capsule contains DCS (237.5 or 175.0 mg) and lurasidone (8.25, 16.5, or 33.0 mg). It is anticipated that subjects entering the study will be receiving concurrent disorder-directed treatment with other approved medications. This treatment regime will be maintained upon entry into the study. However, any use of lurasidone, quetiapine, or olanzapine will be stopped at study entry, so as to avoid either duplication with study drug (groups 1 and 2) or undermining of the control group.

The clinical efficacy goal is to provide extended relief from symptoms associated with Severed Bipolar Depression and ASIB in adults with Bipolar Disorder, after initial stabilization with iv ketamine in a clinic, emergency department, or inpatient setting.

The proposed NRX-101 product takes advantage of a unique synergistic confluence of combining two active pharmaceutical ingredients (DCS and lurasidone) that respectively inhibit the NMDA and the D2/5-HT2A receptors in the brain. NMDA receptor antagonists, most notably ketamine, have been shown in many studies to rapidly reduce depressive and suicidal ideation. However, numerous studies have demonstrated the potential of NMDA antagonists to cause hallucination and other dissociative side effects. Similarly, D2/5HT2A receptor antagonists, such as lurasidone have demonstrated antidepressant effects in bipolar depression, but have demonstrated a propensity to cause akathisia in some patients. The goals of combining these drugs into a single course of treatment is to maximize the beneficial effects of the specific subcomponents while overcoming potential treatment-limiting side effects associated with those subcomponents.

Beneficial effects of the proposed dosage regimen include 1) well-documented pharmacodynamic effects of ketamine in treating both persistent depressive symptoms and suicidal ideation in bipolar disorder (McCloud, 2015; Naughton, 2014; Newport, 2015; Price, 2014), 2) well-documented pharmacodynamic effects of oral DCS against persistent symptoms of depression (Heresco-Levy, 2013) and 3) the FDA-approved efficacy of lurasidone in treatment-resistant depression (Sunovion Pharmaceuticals, 2013). Due to the synergistic effects, the proposed NRX-101 combination capsule is also expected to avoid or minimize the significant undesired adverse effects associated with the usage of these drugs as single agents (eg, negative consequences of repeated use of ketamine (JHP Pharmaceuticals, 2012), potential psychotomimetic effects of long-term treatment with DCS alone (Kantrowitz, 2010) and potential akathisia and susceptibility for increased suicidality associated with lurasidone alone (Sunovion Pharmaceuticals, 2013).

The risk of ASIB is higher in bipolar depression than other psychiatric disorder and the majority of currently available antidepressants are contraindicated for patients with bipolar depression. NeuroRx believes that the proposed NRX-101 treatment regimen (ketamine administration followed by NRX-101) will demonstrate superiority over ketamine followed by lurasidone in maintaining remission from depression and in delaying the time to documented relapse from depression and suicidality in bipolar disorder, providing a new treatment option for patients with Severe Bipolar Depression and ASIB.

There is currently no FDA-approved product for the treatment of ASIB. NeuroRx proposes that NRX-101 will fulfill an urgent medical need for safe and effective treatment for ASIB.

Patients with Severe Bipolar Depression and ASIB will be recruited in inpatient settings and, following informed consent, will be given an intravenous infusion of either ketamine 0.5mg/kg over 40 minutes or normal saline (placebo). Those who exhibit a satisfactory clinical response to ketamine will be randomly allocated to NRX-101 or to lurasidone along (the comparator group). The primary outcome variable for this phase 2 study will be blood level (pharmacokinetic) exposure of NRX-101 and its D-cycloserine component with remission from depression, as measured on the MADRS scale and relapse as secondary endpoints. Relapse is defined as return of either depression or suicidality OR the need to alter therapy, which might include re-hospitalization, additional antidepressant medication, or electroconvulsive therapy (ECT).

ELIGIBILITY:
Inclusion Criteria:A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Male or female, 18 to 65 years of age, inclusive, at screening.
2. Able to read, understand, and provide written, dated informed consent prior to screening. Participants will be deemed likely to comply with study protocol and communicate with study personnel about AEs and other clinically important information.
3. Diagnosed with Bipolar Disorder (BD) according to the criteria defined in the DSM-5. The diagnosis of BD will be made by a site psychiatrist and supported by the MINI 7.0.2. The diagnosis will be confirmed by remote, independent raters, via teleconference between the screen visit and the baseline visit.
4. Suicidal ideation or behavior of sufficient severity to meet the requirements for a score of 4, or 5 on the C-SSRS (suicide attempt, interrupted attempt, aborted attempt, preparatory actions toward imminent suicidal behaviors, active method, intent +/- plan).
5. A score equal to or greater than 20 on the MADRS items of the BISS.
6. In good general health, in the opinion of the investigator, as ascertained by medical history, physical examination (PE) (including measurement of seated vital signs), clinical laboratory evaluations, and electrocardiogram (ECG).
7. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following specific criteria:

   a. Non-childbearing potential (e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized [status post hysterectomy, bilateral tubal ligation], or is post-menopausal with her last menses at least one year prior to screening); or
   * Childbearing potential, and meets the following criteria:

     * Childbearing potential, including women using any form of hormonal birth control, on hormone replacement therapy started prior to 12 months of amenorrhea, using an intrauterine device (IUD), having a monogamous relationship with a partner who has had a vasectomy, or is sexually abstinent.
     * Negative urinary pregnancy test at screening, confirmed by a negative urinary pregnancy test at randomization prior to receiving study treatment.
     * Willing and able to continuously use one of the following methods of birth control during the course of the study, defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly: implants, injectable or patch hormonal contraception, oral contraceptives, IUD, double-barrier contraception, sexual abstinence. The form of birth control will be documented at screening and baseline.
8. Body mass index between 18-35 kg/m2.
9. Concurrent psychotherapy will be allowed if the type (e.g., supportive, cognitive behavioral, insight-oriented) and frequency (e.g., weekly or monthly) of the therapy has been stable for at least three months prior to screening and if the type and frequency of the therapy is expected to remain stable during the course of the subject's participation in the study.
10. Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, benzodiazepines or trazodone) will be allowed if the therapy has been stable for at least 4 weeks prior to screening and if it is expected to remain stable during the course of the subject's participation in the study. Subjects can also continue treatment with benzodiazepines used for sleep or anxiety if therapy has been stable for at least 4 weeks prior to screening and if it is expected to remain stable during the course of the subject's participation in the study.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
2. Female that is pregnant or breastfeeding.
3. Female with a positive pregnancy test at screening or baseline.
4. Current diagnosis of a substance use disorder (abuse or dependence, as defined by DSM-5, with the exception of nicotine dependence), at screening or within 6 months prior to screening.
5. Current Axis I disorder, diagnosed at screening with the use of the MINI 7.0.2, that is the primary focus of treatment and BD the secondary focus of treatment for the past 6 months or more.
6. History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms.
7. History of anorexia nervosa, bulimia nervosa, or eating disorder not otherwise specified, within 5 years of screening.
8. Any Axis I or Axis II Disorder, which at screening is clinically predominant to their BD or has been predominant to their BD at any time within 6 months prior to screening.
9. Has dementia, delirium, amnestic, or any other cognitive disorder.
10. Has a clinically significant abnormality on the screening physical examination that might affect safety, study participation, or confound interpretation of study results according to the study clinician.
11. Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation.
12. Current episode of:

    * Hypertension, Stage 1 as defined by a systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg at screening on two of three measurements at least 15 minutes apart.
    * Hypertension, Stage 1 as defined by a systolic blood pressure ≥155 mmHg or diastolic blood pressure ≥99 mmHg at the Baseline Visit (Visit 1) within 1.5 hours prior to ketamine infusion on two of three measurements at least 15 minutes apart.
    * Recent myocardial infarction (within one year) or a history of myocardial infarction.
    * Syncopal event within the past year.
    * Congestive heart failure (CHF) New York Heart Association Criteria >Stage 2
    * Angina pectoris.
    * Heart rate <50 or >105 beats per minute at screening or randomization (Baseline Visit).
    * QTcF (Fridericia-corrected) ≥450 msec at screening or randomization (Baseline Visit).
13. Current history of hypertension, or on antihypertensives for the purpose of lowering blood pressure, with either an increase in antihypertensive dose or increase in the number of antihypertensive drugs used to treat hypertension over the last 2 months.
14. Chronic lung disease excluding asthma.
15. Lifetime history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention which, according to the screening clinician, is deemed associated with significant injury to or malfunction of the CNS, or history of significant head trauma within the past 2 years.
16. Presents with any of the following lab abnormalities:

    * Subjects with diabetes mellitus fulfilling any of the following criteria:

      * Unstable diabetes mellitus defined as glycosylated hemoglobin (HbA1c) >8.5% at screening.
      * Admitted to hospital for treatment of diabetes mellitus or diabetes mellitus-related illness in the past 12 weeks.
      * Not under physician care for diabetes mellitus.
      * Has not been on the same dose of oral hypoglycemic drug(s) and/or diet for the 4 weeks prior to screening. For thiazolidinediones (glitazones) this period should not be less than 8 weeks.
    * Any other clinically significant abnormal laboratory result (determined as such by the investigator and medical monitor) at the time of the screening.
17. Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.
18. Positive screening urine test for drugs of abuse at screening: cocaine, amphetamines, barbiturates, opiates.
19. Subjects with exclusionary laboratory values, or requiring treatment with exclusionary concomitant medications as defined in the study manual
20. Subjects on exclusionary concomitant psychotropic medications.
21. Subjects with a lifetime history of illicit PCP/ketamine drug use or previous failed use of ketamine for depression.
22. Liver Function Tests higher than 2.5 times upper limit of normal as defined in the study manual.
23. Known allergies to Lurasidone or Latuda, Cycloserine or Seromycin, Mannitol, Croscarmellose Sodium, Magnesium Stearate, Silicon Dioxide, and/or HPMC (hydroxypropylmethylcellulose)

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Nierenberg, MD, Principal Investigator — Massachusetts General Hospital; Daniel C Javitt, MD, Study Director — NeuroRx, Inc.
Locations (4):
- United States (4):
  - Research Site, Birmingham, Birmingham, Alabama
  - Research Site, Fort Lauderdale, Fort Lauderdale, Florida
  - Research Site, Charlotte, Charlotte, North Carolina
  - Research Site, Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nierenberg A, Lavin P, Javitt DC, Shelton R, Sapko MT, Mathew S, Besthof RE, Javitt JC. NRX-101 (D-cycloserine plus lurasidone) vs. lurasidone for the maintenance of initial stabilization after ketamine in patients with severe bipolar depression with acute suicidal ideation and behavior: a randomized prospective phase 2 trial. Int J Bipolar Disord. 2023 Aug 13;11(1):28. doi: 10.1186/s40345-023-00308-5. PMID 37573534

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine Followed by NRX-101: NRX-101 is a fixed dose combination of d-cycloserine and lurasidone
  NRX-101 Oral Capsule: Prospective Randomized Factorial Design Study as per arm/group descriptions
  Ketamine Intravenous Infusion: Randomized administration of Ketamine or Placebo in a 3 to 1 ratio
  Saline Solution Intravenous Infusion: Randomized administration of Ketamine or Placebo in a 3 to 1 ratio
- Ketamine Followed by Lurasidone: Lurasidone will be administered in the same dosages as the lurasidone component of NRX-101
  Lurasidone Oral Capsule: Prospective Randomized Factorial Design Study as per arm/group descriptions
  Ketamine Intravenous Infusion: Randomized administration of Ketamine or Placebo in a 3 to 1 ratio
  Saline Solution Intravenous Infusion: Randomized administration of Ketamine or Placebo in a 3 to 1 ratio
- Saline Followed by NRX-101; Saline Followed by Lurasidone: Lurasidone will be administered in the same dosages as the lurasidone component of NRX-101
  Lurasidone Oral Capsule: Prospective Randomized Factorial Design Study as per arm/group descriptions
  Saline Solution Intravenous Infusion: Randomized administration of Ketamine or Placebo in a 3 to 1 ratio
Period: Overall Study
Arm/Group | Ketamine Followed by NRX-101 | Ketamine Followed by Lurasidone | Saline Followed by NRX-101 | Saline Followed by Lurasidone
Started | 12 | 5 | 4 | 1
Completed | 6 | 2 | 2 | 1
Not Completed | 6 | 3 | 2 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Completed day 42 but did not return for day 70 | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ketamine Followed by NRX-101: NRX-101 is a fixed-dose combination of d-cycloserine and lurasidone
  NRX-101 Oral Capsule: Prospective Randomized Factorial Design Study as per arm/group descriptions
  Ketamine Intravenous Infusion: Randomized administration of Ketamine or Placebo in a 3 to 1 ratio
  Saline Solution Intravenous Infusion: Randomized administration of Ketamine or Placebo in a 3 to 1 ratio
- Saline Followed by NRX-101; Saline Followed by Lurasidone: Lurasidone will be administered in the same dosages as the lurasidone component of NRX-101
  Lurasidone Oral Capsule: Prospective Randomized Factorial Design Study as per arm/group descriptions
  Ketamine Intravenous Infusion: Randomized administration of Ketamine or Placebo in a 3 to 1 ratio
  Saline Solution Intravenous Infusion: Randomized administration of Ketamine or Placebo in a 3 to 1 ratio
- Total: Total of all reporting groups
Arm/Group | Ketamine Followed by NRX-101 | Ketamine Followed by Lurasidone | Saline Followed by NRX-101 | Saline Followed by Lurasidone | Total
Number analyzed (Participants) | 12 | 5 | 4 | 1 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (10.5) | 49 (8.9) | 41 (8.9) | 54 (0) | 39.5 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 2 | 1 | 16
  Male | 3 | 1 | 2 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 11 | 5 | 3 | 0 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 5 | 4 | 1 | 22
Columbia Suicide Severity Rating Scale (CSSRS) [Number; unit: participants] — Columbia Suicide Severity Rating Scale (C-SSRS): C-SSRS is a well validated, low-burden measure of the spectrum of suicidal ideation and behavior that was developed in the National Institute of Mental Health Treatment of Adolescent Suicide Attempters Study to assess severity and track suicidal events through any treatment. . It contains a 1-to-5 rating scale for suicidal ideation of increasing severity (from a "wish list to die" to an "active thought of killing oneself with plan and intent").
  participants
    CSSRS = 1 | 1 | 0 | 0 | 0 | 1
    CSSRS = 2 | 0 | 0 | 0 | 0 | 0
    CSSRS =3 | 0 | 0 | 0 | 0 | 0
    CSSRS =4 | 2 | 0 | 0 | 0 | 2
    CSSRS = 5 | 9 | 5 | 4 | 1 | 19

OUTCOME MEASURES:

1. Primary Outcome: BDM Score (BISS-derived MADRS) Change From Baseline at Day 42
Description: The study will measure the difference on BISS-derived MADRS score between NRX-101 and lurasidone (comparator) groups. The Bipolar Inventory of Symptom Scale (BISS) is a validated 42-item clinician-rated scale (21 items each for the depression and mania subscales) in which each item is rated on a 0-4 severity scale where higher values indicate worse severity.
  BISS-derived MADRS (BDM): MADRS is a 10-item clinician-rated scale, with each item rated on a 0-6 severity scale, where a higher number indicates worse severity. Responses to each question are equally weighted and summed. The BDM has a minimum score of 0 and a maximum of 40, where higher scores indicate a worse severity, therefore decreases in average BDM are considered a better outcome. Data are presented as mean change from baseline (end of stage 1, Day 1) using LOCF
Time Frame: Day 42
Population: Last Observation Carrier Forward
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Saline Followed by NRX-101: Saline (stage 1) followed by NRX-101 (stage 2)
- Saline Followed by Lurasidone: Saline (stage 1) followed by lurasidone (stage 2)
Arm/Group | Ketamine Followed by NRX-101 | Ketamine Followed by Lurasidone | Saline Followed by NRX-101 | Saline Followed by Lurasidone
Number analyzed (Participants) | 12 | 5 | 4 | 1
score on a scale
  Day 2 | 3.3 (1.95) | 2.4 (2.95) | -1.06 (3.81) | 0 (0)
  Day 7 | 2.0 (1.91) | 4.8 (2.95) | -0.5 (3.74) | 0 (0)
  Day 14 | 2.2 (1.91) | 11.4 (2.95) | 0.31 (4.0) | 0 (0)
  Day 21 | 4.5 (1.91) | 10.0 (2.95) | 1.0 (5.72) | 0 (0)
  Day 28 | 3.5 (1.91) | 11.2 (2.95) | 1.69 (7.34) | 0 (0)
  Day 35 | 2.8 (1.91) | 10.8 (2.95) | 1.75 (8.43) | 0 (0)
  Day 42 | 3.7 (1.91) | 11.0 (2.95) | 0.38 (5.77) | 0 (0)
Statistical Analysis 1: Comparison: Ketamine Followed by NRX-101 vs Ketamine Followed by Lurasidone; Test type: Superiority; p = .03, Mixed Models Analysis — BDM LS difference overall; BDM LS difference overall

ADVERSE EVENTS:
Time Frame: Study Duration (6 weeks)
Arm/Group | Ketamine Followed by NRX-101 | Ketamine Followed by Lurasidone | Saline Followed by NRX-101 | Saline Followed by Lurasidone
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/5 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/5 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 8/12 | 3/5 | 4/4 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine Followed by NRX-101 (N=12) | Ketamine Followed by Lurasidone (N=5) | Saline Followed by NRX-101 (N=4) | Saline Followed by Lurasidone (N=1)
tinnitus (Ear and labyrinth disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
dysmetropsia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypoasthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dissociation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
euphoric mood (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
restlessness (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vision blurred (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
abdominal distention (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
fatigue (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
thermal burn (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
akathisia (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
sedation (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
anorgasmia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
restlessness (Psychiatric disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ejaculation delayed (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT02974010/Prot_SAP_000.pdf